CLINICAL TRIAL: NCT05494814
Title: Sandhills Central Community Kitchen Evaluation: Using the Veggie Meter
Brief Title: Sandhills Community Kitchen Evaluation: Using the Veggie Meter
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The central kitchen, designed to prepare and serve meals to child care centers, that this study was designed to evaluate, never launched its business.
Sponsor: North Carolina State University (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Jessica Bloom, Associate Professor and Local Foods Extension Specialist, North Carolina State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24444
Record Dates: First submitted 2022-04-27; First posted 2022-08-10 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Diet, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Child Care Centers Served Meals Prepared by Central Kitchen (Experimental): Children ages 3-5 attending a child care center that purchases meals prepared by a central kitchen.
  Interventions: Other: Child Care Centers Served Meals Prepared by Central Kitchen
- Child Care Centers Not Served Meals Prepared by Central Kitchen (No Intervention): Children ages 3-5 attending a child care center that does not purchase meals prepared by a central kitchen.

INTERVENTIONS:
Other: Child Care Centers Served Meals Prepared by Central Kitchen — The child care centers who are served by the central kitchen will receive meals that include locally sourced fresh fruits and vegetables to serve their staff and children.
  Arms: Child Care Centers Served Meals Prepared by Central Kitchen

SUMMARY:
This clinical trial will evaluate the development, implementation, and impact of a central kitchen preparing and serving meals to child care centers in rural Harnett County, North Carolina. The goals of the kitchen are to improve meal quality, reduce workload on child care providers, create a sustainable business model, and provide a source of community economic development. Our evaluation of the Sandhills Central Community Kitchen is important to better understand how this model can be replicated to serve rural communities. We will recruit 20 child care centers (10 intervention and 10 as a control group); we estimate that each child care center will serve 40 children. We will collect baseline data at the beginning of the project from all 20 centers, and will repeat data collection at the end of the project to assess changes. Data will be collected through parent surveys, surveys and interviews with child care center directors, surveys and focus groups with teachers, interviews with the church pastor and community leaders where the kitchen is based, surveys of kitchen staff, nutritional analysis of menu data, collection and analysis of food costs, and through use of the "Veggie Meter" (a non-invasive instrument that assesses changes in intake of fruits and vegetables by measuring skin carotenoids) with child care center children and staff. Our goal is to document the impacts of central kitchens in terms of nutritional and economic benefits in order to create a replicable model.

DETAILED DESCRIPTION:
This clinical trial will evaluate the development, implementation, and impact of a central kitchen preparing and serving meals to child care centers in rural Harnett County, North Carolina. The goals of the kitchen are to improve meal quality, reduce workload on child care providers, create a sustainable business model, and provide a source of community economic development. Our evaluation of the Sandhills Central Community Kitchen is important to better understand how this model can be replicated to serve rural communities. We will recruit 20 child care centers (10 intervention and 10 as a control group); we estimate that each child care center will serve 40 children. We will collect baseline data at the beginning of the project from all 20 centers, and will repeat data collection at the end of the project to assess changes. Data will be collected through parent surveys, surveys and interviews with child care center directors, surveys and focus groups with teachers, interviews with the church pastor and community leaders where the kitchen is based, surveys of kitchen staff, nutritional analysis of menu data, collection and analysis of food costs, and through use of the "Veggie Meter" (a non-invasive instrument that assesses changes in intake of fruits and vegetables by measuring skin carotenoids) with child care center children and staff. Our goal is to document the impacts of central kitchens in terms of nutritional and economic benefits in order to create a replicable model.

Skin carotenoid status (SCS) will be used to measure F&V intake among pre-schoolers. Carotenoids, the colorful phytonutrients found in vegetables are correlated with F&V intake. A higher carotenoid level is correlated with higher F&V intake; conversely lower carotenoid levels are associated with lower F&V intake over the past month. To measure carotenoid level, researchers will use the Veggie Meter®. The Veggie Meter is a small, portable, non-invasive device that assesses SCS via pressure-mediated reflection spectroscopy. This is more accurate than self-reported diet among children.

ELIGIBILITY:
Inclusion Criteria: Must be a child enrolled at a child care center that purchases meals from a central kitchen.

-

Exclusion Criteria: No exclusion criteria.

-

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in produce intake | Will be assessed pre-intervention and one year later.
  Measured through "Veggie Meter" scans of child care center children and staff, which measure the level of carotenoids in the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Dara Bloom, PhD, Principal Investigator — North Carolina State University
Locations (1):
- North Carolina State University, Raleigh, North Carolina, United States